CLINICAL TRIAL: NCT01224873
Title: Diagnosis of Sceletal Metastases in c. Mammae: 18F-NaF-PET/Lowdose-CT Versus 99mTc HDP Bone Scintigraphy
Brief Title: Diagnosis of Bone Metastases in Breast Cancer: Bone Scintigraphy, Fluoride-PET and FDG-PET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Dr. Christine Winkler, Department of Nuclear Medicine & PET
Other Study IDs: H-3-2010-019
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; bone metastasis; comparison of diagnostic methods; bone scintigraphy; fluoride PET/CT; FDG-PET/CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Breast cancer can metastasize to the bones, which leads to another treatment if bone metastases are detected. The purpose of the study is to determine, if fluoride PET/CT is superior to bone scintigraphy with technetium. On the other side, the investigators would like to see if FDG-PET/CT is a reliable alternative to dedicated bone imaging to detect bone metastases in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven c. mammae
* clinically suspicion of bone metastases

Exclusion Criteria:

* age under 18 years
* diabetes mellitus
* pregnancy
* other known malignant disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients who are treated at Rigshospitalet, DK
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Winkler, Dr., Principal Investigator — Dep. of Nuclear Medicine & PET, Rigshospitalet, Denmark
Locations (1):
- Dep. of Nuclear Medicine & PET, Rigshospitalet, Copenhagen, Denmark